CLINICAL TRIAL: NCT06955767
Title: Performance of Serum Matrix Metalloproteinase (MMP14) Assay as a Novel Biomarker for Colorectal Cancer Screening in Subjects From 50 to 74 Years Old Referred for Colonoscopy After Positive FIT
Brief Title: Measurement of MMP-14 Protein, a Potential New Marker for Colorectal Cancer Detection, in Plasma Vesicles Named Exosomes
Acronym: EXOSCOL02
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PR25047
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Adenocarcinoma
Keywords: Colorectal Adenocarcinoma; Exosomes; Matrix Metalloproteinase 14; MMP-14

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serum Matrix Metalloproteinase (MMP14) (Experimental): Blood will be drawn from 2 additional tubes of 5 ml each, either in the consultation room or in the operating room.
  Interventions: Other: Blood will be drawn from 2 additional tubes of 5 ml each

INTERVENTIONS:
Other: Blood will be drawn from 2 additional tubes of 5 ml each — Blood will be drawn from 2 additional tubes of 5 ml each

SUMMARY:
Colorectal cancer is the third most common cancer in men, and the second most common in women. Screening for colorectal cancer is based on the search for blood in the stool using fecal immunochemical test (FIT). Occult bleeding is an indication for colonoscopy. In a FIT positive population, 60% of colonoscopies are negative, 34% diagnose an adenomatous lesion, and 6% a cancer. The identification of new biological markers could reduce the number of colonoscopies performed. Cancer cells release extracellular vesicles that contain proteins, mRNAs, DNA, which they can transfer to neighbouring or distant cells. The use of exosomal proteins as novel tumor markers looks very promising. We performed a pilot study comparing the levels of different exosomal proteins in 74 subjects which was recently accepted for publication in Journal of Clinical Laboratory Analysis. Comparison of results showed that only matrix metalloproteinase 14 (MMP14) was significantly higher in patients with colorectal cancer or adenoma than in people with normal colonoscopy.

The primary objective of the current study is to determine the best cut-off value of MMP-14 for colorectal cancer screening and to evaluate the performance (Sensitivity, Specificity…) associated to this cut-off value. The secondary objective will be to determine the best cut-off value of MMP-14 for colorectal adenomas screening and to evaluate its performance.

For this purpose, 650 patients, seen for diagnostic colonoscopy following a positive FIT test, will be included in the study. After blood collection and exosome isolation, MMP-14 will be measured using a quantitative test (enzyme-linked immunosorbent assay) and the results will be associated with colonoscopy results to determine the sensitivity, specificity, positive predictive value (PPV) and net present value (NPV).

DETAILED DESCRIPTION:
Inclusion criteria: Individuals presenting for colonoscopy with a positive FIT result.

* Positive fecal immunoassay requiring total colonoscopy under general anesthesia.
* Persons having agreed to participate in the study (signed consent form)
* Adults affiliated to a health insurance scheme.

Non-inclusion criteria:

* History of other cancer not in remission or in remission for less than five years (with the exception of cervical cancer or basal cell skin cancer treated with curative intent)
* Patients undergoing chemotherapy
* Patients protected by law This is a cross-sectional multicenter interventional study. Patients will be recruited from the Hepato-Gastroenterology departments of the CHU de Reims, CHU de Dijon, CHU de Nancy, CHU de Besançon, CH de Châlons-en-Champagne, Institut Jean Godinot de Reims, CHU de Strasbourg, CH de Charleville Mézières and CH d'Epernay.

Once consent has been signed and the patient has been included in the study, blood will be drawn from 2 additional tubes of 5 ml each, either in the consultation room or in the operating room, when the infusion is set up for colonoscopy under general anaesthetic. Plasma will be collected at the various participating facilities (2 x 5mL EDTA tubes), centrifuged at 1000g for 10 minutes, then frozen at -80°C. Samples will then be sent to the Reims University Hospital Biology Department for storage before analysis.

The isolation of exosomes from the patient's plasma and their characterization: size, number (determined using the Malvern Panalytical NanoSight NS300), and MMP14 concentration (determined by enzyme-linked immunosorbent assay), will be carried out at the CNRS UMR7369 "Matrice Extracellulaire et Dynamique Cellulaire (MEDyC)" unit at the University of Reims Champagne Ardenne.

ELIGIBILITY:
Inclusion criteria:

* Individuals presenting for colonoscopy with a positive FIT result.
* Positive fecal immunoassay requiring total colonoscopy under general anesthesia.
* Persons having agreed to participate in the study (signed consent form)
* Adults affiliated to a health insurance scheme.

Exclusion criteria:

* History of other cancer not in remission or in remission for less than five years (with the exception of cervical cancer or basal cell skin cancer treated with curative intent)
* Patients undergoing chemotherapy
* Legally protected individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Serum Matrix Metalloproteinase (MMP14) : normal versus a cancerous lesion | At 30 minutes
  Concentration of Serum Matrix Metalloproteinase (MMP14) depending on whether the colonoscopy was normal or revealed a cancerous lesion

SECONDARY OUTCOMES:
Serum Matrix Metalloproteinase (MMP14) MMP14 Concentration: Normal vs. Adenoma | At 30 minutes
  Concentration of Serum Matrix Metalloproteinase (MMP14) depending on whether the colonoscopy was normal or revealed an adenoma
Serum MMP14 Concentration according to adenoma characteristics | At 30 minutes
  Concentration of Serum Matrix Metalloproteinase (MMP14) according to adenoma characteristics
Serum MMP14 Concentration between groups: normal colonoscopy vs. adenoma and cancerous lesions | At 30 minutes
  Comparison of exosomal plasma MMP14 concentration between groups: normal colonoscopy vs. adenoma and cancerous lesions
Diagnostic performances of Serum MMP14 | At 30 minutes
  Sensitivity and specificity
Concentration of markers derived from circulating tumor exosomes in the context of colorectal cancer | At 30 minutes
  Mean value of markers derived from circulating tumor exosomes

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France